CLINICAL TRIAL: NCT06285890
Title: Phase I Study of HC-7366 for Acute Myeloid Leukemia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: HiberCell, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-1016; NCI-2024-01733 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): If you are found to be eligible to take part in this study, you will be assigned to a dose level of HC-7366 based on when you join this study. Participants enrolled will receive HC-3766 single agent. HC-3766 will be taken once daily while fasting, 1 hour before or 2 hours after a meal, on days 1-28.
  Interventions: Drug: HC-7366

INTERVENTIONS:
Drug: HC-7366 — Given by PO

SUMMARY:
To find a recommended dose of HC-7366 to patients with AML. The safety and effects of this drug combination will also be studied.

DETAILED DESCRIPTION:
Primary Objective:

- To evaluate safety of HC-7366

Secondary Objectives:

* To estimate rate of CR/CRh/CRi by 4 cycles
* To estimate overall response rate (ORR)
* To estimate rate of MRD negative by 4 cycles
* To estimate overall survival (OS)
* To estimate relapse-free survival (RFS)

Exploratory Objectives

* To determine the plasma concentration and pharmacokinetic (PK) parameters of HC-7366 when dosed in combination with azole antifungals in AML patients.
* To estimate duration of response (DOR)
* To estimate median time to blood count recovery
* To estimate median time to first response
* To estimate median time to negative MRD
* To study drug-drug interactions with CYP3A4 inhibitor azole antifungals
* Additional response and survival endpoints.
* To explore biomarkers of response, pathway engagement, and resistance

ELIGIBILITY:
Inclusion Criteria:

1. Patients need to have a confirmed diagnosis of AML, or MDS/AML with 10% to 19% blasts, per the International Consensus Classification 2022 or the WHO 2022 classification.

   Dose escalation phase
2. Patients ≥18 years with R/R AML or R/R MDS/AML, other than acute promyelocytic leukemia (APL), with no available standard treatment options.
3. Relapsed or refractory disease defined by standard criteria as follows:

   a. Relapsed: Bone marrow blasts ≥5%, reappearance of blasts in the blood, or development of extramedullary disease following achievement of CR/CRi/MLFS b. Refractory: Failure to achieve CR/CRi/MLFS following initial treatment, with evidence of persistent leukemia by blood and/or bone marrow evaluation with blasts ≥5% c. Appropriate prior therapy in order for patient to be deemed relapsed or refractory include any of the following: i. At least 1 cycle of purine analogue containing intensive induction chemotherapy regimen, e.g., FLAG-Ida, CLIA or CLAG-M or similar regimens with or without venetoclax.

   ii. At least 1 cycle of intensive induction chemotherapy with venetoclax, e.g., 7 + 3 or CPX-251 with venetoclax or similar regimens iii. At least 2 cycles of intensive induction chemotherapy such as 7 + 3 or 5 + 2 or similar regimens without venetoclax iv. 2 cycles of venetoclax with HMA/LDAC +/- other agents v. 4 cycles of HMA alone d. Younger/fit patients in first relapse following intensive chemotherapy, will only be eligible if the first remission (CR1) duration was ≤12 months.

   e. Participants relapsing with persistent or new TP53 mutation will be eligible irrespective of CR1 duration.

   f. Older/unfit patients who relapse on HMA + venetoclax based maintenance regimen will be eligible irrespective of CR1 duration
4. ECOG PS 0 to 2
5. Patients relapsing after allo-SCT may be eligible if they have recovered from all transplantrelated toxicities and are off all immunosuppression, with no more than grade 1 chronic GVHD. Physiologic ("replacement") dose of steroids (≤10 mg prednisone or equivalent) may be acceptable. Patients must be off all immunosuppression, including calcineurin inhibitors, for at least 2 weeks or 5 half-lives, whichever is longer, prior to enrollment on study.
6. Patients with actionable mutations with available FDA-approved therapies, e.g., FLT3, IDH1/2 inhibitors may be enrolled after they have exhausted appropriate lines of FDA approved treatment options.
7. Patients with antecedent hematological disorder (AHD), e.g., aplastic anemia, myelodysplastic syndrome (MDS), chronic myelomonocytic leukemia (CMML) or myeloproliferative disorder or neoplasm (MPD or MPN) who have previously received a regimen appropriate for AML for the antecedent hematological disorder, as described above, and have progressed to AML, will be eligible for the dose escalation phase. This is due to recognized poor outcomes in such patients with "treated secondary AML".

   All Participants
8. Adequate hepatic function (total bilirubin ≤1.5 x upper limit of normal (ULN) unless increase is due to Gilberts's disease or leukemic involvement, and AST and/or ALT ≤ 2.5 x ULN unless considered due to leukemic involvement, in which case total bilirubin or AST and/or ALT ≤ 3 x ULN will be considered eligible).
9. Adequate renal function with creatinine clearance ≥ 45 mL/min calculated by the Cockcroft-Gault formula or MDRD equation or measured by 24-hour urine collection.
10. The effects of these agents on the developing human fetus are unknown. For this reason, and because other therapeutic agents used in this trial may be teratogenic, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 90 days after last treatment.

    a. This includes all female participants between the onset of menses (as early as 8 years of age) and 55 years unless the patient presents with an applicable exclusionary factor which may be one of the following: i. Postmenopausal (no menses in greater than or equal to 12 consecutive months).

    ii. History of hysterectomy or bilateral salpingo-oophorectomy. iii. Ovarian failure (follicle-stimulating hormone and estradiol in menopausal range, who have received whole pelvic radiation therapy).

    iv. History of bilateral tubal ligation or another surgical sterilization procedure.

    b. Approved methods of birth control are as follows: Hormonal contraception (i.e., birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), tubal ligation or hysterectomy, subject/partner post vasectomy, implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however, periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.

    c. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of treatment.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients with t(15;17) karyotypic abnormality.
2. Patient has a white blood cell count > 15 x 10⁹/L. Hydroxyurea, and/or cytarabine (up to 2 g/m2 total) used as supportive care is permitted to meet this criterion.
3. Prior use of any cytotoxic chemotherapy, targeted therapy, radiation therapy, immunotherapy, or other clinical trial therapies within 2 weeks, prior to first dose of study treatment. Patients should have recovered from all prior therapy related toxicities. Patients may receive hydroxyurea or cytarabine for control of WBC count during this washout period.
4. Patients with known symptomatic or uncontrolled CNS leukemia.
5. Patient has systemic fungal, bacterial, viral or other infection that is exhibiting ongoing signs/symptoms related to the infection without improvement despite appropriate treatment.
6. Patients with any severe gastrointestinal or metabolic condition which could interfere with absorption of oral study medications or history of chronic diarrhea, enteritis, colitis, inflammatory bowel disease, irritable bowel syndrome. Patients with remote history of such events may be allowed based on review and discussion with PI.
7. Active and uncontrolled comorbidities including decompensated congestive heart failure NYHA class III/IV, clinically significant, uncontrolled arrhythmia, acute respiratory failure, unstable or decompensated pulmonary disease, as judged by the treating physician.
8. Known active hepatitis B (HBV) or Hepatitis C (HCV) infection with detectable viral DNA or RNA, respectively, or known HIV infection.
9. Decompensated congestive heart failure, hypokalemia, prolonged QT interval corrected for heart rate (QTc) (as calculated using Fridericia's formula) to greater than 450 msec for males, or to greater than 470 msec for females or long QT syndrome, or history of Torsades de pointes. Patients with bundle branch block or pacemaker and prolonged QTc interval are permitted after appropriate correction, (e.g., Bogossian formula, or others) or after discussion with the PI and/or cardiologist.

11. Any previous malignancy, except when the patient has completed definitive curative-intent treatment with chemotherapy and/or surgery and/or radiotherapy at least 1 month prior to enrollment. Patients having completed definitive treatment for the following conditions may be eligible immediately after completion of definitive curative-intent therapy, after healing of wounds, and no evidence of residual disease by examination or imaging or cytology/pathology, e.g., non-melanoma skin cancers, or any carcinoma in-situ, e.g., ductal carcinoma in situ, urothelial cancer, cervical cancer, localized prostate cancer, pre-cancerous colon polyp, etc.

12. Major surgery within 4 weeks prior to screening or a major wound that has not fully healed.

13. Patients under legal protection measure (guardianship, trusteeship or safeguard of justice) and/or uncontrolled psychiatric comorbidities, ongoing illicit substance abuse, inability, any impairment or unwillingness to comply with the treatments, follow-up, requirements and procedures of this clinical trial.

14. A known hypersensitivity or severe allergy to study drug components or diluents.

15. Nursing women, women of childbearing potential (WOCBP) with positive urine or serum pregnancy test, or WOCBP who are not willing to maintain adequate contraception.

16. Pregnant women are excluded from this study because study agents may have the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with study agents, breastfeeding should be discontinued if the mother is treated on this study.

17. The study will exclude first-degree relatives of the investigator, study staff or industry sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Abhishek Maiti, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org